CLINICAL TRIAL: NCT05920928
Title: Comparison of the Clinical Response of Total nEoadjuvant Treatment of Two Methods of Long-term or Short-term cHemoRadiotherapy Followed by Consolidation Chemotherapy in Patients With Locally Advanced rectAl Cancer (TEHRAN) , a Randomized Controlled Clinical Trial
Brief Title: Comparison of the Clinical Response of Total Neoadjuvant Treatment of Two Methods of Long-term or Short-term Chemoradiotherapy in Rectal Cancer
Acronym: TEHRAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.TUMS.IKHC.REC. 9911880002
Record Dates: First submitted 2023-06-05; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Locally Advanced Rectal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Long course chemoRadiotherapy (50.4Gy in 28 fr) (Experimental): Neoadjuvant Long course radiotherapy (50.4 Gy in 28 fr) with concurrent capecitabine (825mg/m2) for locally advanced rectal cancer
  Interventions: Radiation: Long course radiotherapy with concurrent capecitabine(825mg/m2)
- Short course chemoRadiotherapy (25Gy in 5 fr) (Experimental): Neoadjuvant short course radiotherapy (25 Gy in 5 fr) with concurrent capecitabine (825mg/m2) for locally advanced rectal cancer
  Interventions: Radiation: Short course radiotherapy with concurrent capecitabine(825mg/m2)

INTERVENTIONS:
Radiation: Short course radiotherapy with concurrent capecitabine(825mg/m2) — Compared to conventional treatments, short-term radiotherapy has lower fraction numbers but higher radiation doses per fraction. capecitabine is given during treatment time (825mg/m2)
  Other Names: Short term radiotherapy (25Gy in 5Fr)
  Arms: Short course chemoRadiotherapy (25Gy in 5 fr)
Radiation: Long course radiotherapy with concurrent capecitabine(825mg/m2) — Long-term radiation is administered in conjunction with concomitant capecitabine (825mg/m2)
  Other Names: Long term radiotherapy (50.4Gy in 28Fr)
  Arms: Long course chemoRadiotherapy (50.4Gy in 28 fr)

SUMMARY:
Rectal cancer is one of the most prevalent malignancies in the world, and its prevalence is rising. In more advanced cases neoadjuvant therapy is advised before to surgery, and radiotherapy is one of its cornerstones. For the treatment of rectal cancer, there are primarily two radiation techniques. Long-term radiotherapy is 50.4 Gy delivered in 28 fractions, while short-term radiotherapy is 25 Gy delivered in 5 parts. In earlier studies, these two radiation techniques were combined with various chemotherapy drugs, and a relative comparison was established. Total neoadjuvant treatment, or TNT, has been linked to a better outcome because of the significance of organ preservation. The aim of this research is to compare two TNT radiation techniques with the same regimen of treatment.

ELIGIBILITY:
Inclusion Criteria:

Locally advanced (T3-4, N+)adenocarcinoma of rectum that is located 5 to 15 cm from anal verge .

Exclusion Criteria:

Familial syndromes e.g. lynch Previous history of cancer Previous history of chemotherapy Recurrent disease Metastatic disease Inability to perform MRI (Claustrophobia or prosthetic valve)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-09-23 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response | Week
  At the 18th week following the start of the treatment, the patient will be assessed. The evaluation consist of an MRI and a colonoscopy, with a PET scan being optional.

REFERENCES:
- [Derived] Aghili M, Ghalehtaki R, Yaghooti-Khorasani M, Yazdi SMM, Kolahdouzan K. Comparison of the Clinical Response in Total Neoadjuvant Treatment With Long-Term or Short-Term Chemoradiotherapy Followed by Consolidation Chemotherapy in Patients With Locally Advanced Rectal Cancer (TEHRAN); the Protocol for a Randomized Controlled Clinical Trial. Cancer Med. 2025 Dec;14(24):e71472. doi: 10.1002/cam4.71472. PMID 41412957